CLINICAL TRIAL: NCT06370702
Title: Evaluating the Use of Grip Exercises to Decrease Deep Vein Thrombosis in Adult Patients With PICC Lines
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-054
Record Dates: First submitted 2023-12-19; First posted 2024-04-17 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handgrip Exercise Group (Experimental): Participants will be instructed to firmly grip and squeeze the ball for 10 seconds, relax for 10 seconds and repeat for 10 minutes. They will be instructed to do this 3 times per day.
  Interventions: Other: Handgrip Exercises
- Standard Care Group (No Intervention): Participants will receive standard care that includes no instruction about conducting hand grip exercises.

INTERVENTIONS:
Other: Handgrip Exercises — Participants will firmly grip and squeeze the ball for 10 seconds, relax for 10 seconds and repeat for 10 minutes. They will be instructed to do this 3 times per day.
  Arms: Handgrip Exercise Group

SUMMARY:
Patients who have a peripherally-inserted central catheter (PICC) placed are at a risk of developing a deep vein thrombosis (DVT). At TriHealth, approximately 2-4 patients per month who have a PICC placed experience a subsequent DVT. One innovative way to possibly mitigate the risk of DVTs is hand grip exercises. The current study will be the first study to evaluate hand grip exercises for the prevention of DVTs in adult patients hospitalized in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Had a PICC placed in the past 24 hours by the Vascular Access Team
* Patient is admitted to either Bethesda North Hospital or Good Samarian Hospital

Exclusion Criteria:

* Under 18 years old
* Does not speak English
* Unable to consent to involvement in the research study
* Has a bleeding disorder/diagnosis
* Has a severe limb disfunction whereby they would be unable to perform the grip exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Deep vein thrombosis | from PICC placement to PICC removal, up to 4 weeks
  Incidence of deep vein thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Baker, PhD, RN, Study Chair — TriHealth Nurse Researcher
Locations (2):
- United States (2):
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No